CLINICAL TRIAL: NCT00527722
Title: A Prospective Randomized Multi-Centered Study and Efficacy Evaluation of the Bio-Seal Biopsy Track Plug for Reducing Pneumothorax Rates Post Lung Biopsy Procedures
Brief Title: Evaluation of the Bio-Seal Biopsy Track Plug
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2005-0268
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Bio-Seal Track Plug; Lung Biopsy; Lung Plug; Air Leaks
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pleural Plug (Experimental): Experimental lung plug after the lung biopsy.
  Interventions: Device: Bio-Seal Track Plug
- No Pleural Plug (Active Comparator): The standard lung biopsy without placement of the plug.
  Interventions: Other: No lung plug

INTERVENTIONS:
Device: Bio-Seal Track Plug — The lung plug will be inserted into the left track when the biopsy needle is removed. The smaller sampling needle is removed, and the lung plug is inserted through the larger needle using a delivery tool that has a plunger to push the plug in place. The lung plug remains in the track left when the larger needle is removed.
  Arms: Pleural Plug
Other: No lung plug — Standard lung biopsy without placement of the plug.
  Arms: No Pleural Plug

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the Bio-Seal Biopsy Track Plug in a clinical setting for use in lung biopsy procedures to reduce the rate of air leaks, commonly associated with the procedure. The Bio-Seal System is cleared in the U.S. with an indication for use as a lung biopsy site marker.

DETAILED DESCRIPTION:
Air leaks are the most common problem after a lung biopsy. Air leaks can be mild to severe. Mild air leaks are monitored by chest x-ray and may go away by themselves. Air leaks can cause pain and require repeated x-rays, and in some cases the need for a tube to be inserted into the chest for drainage of the air.

If you agree to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1of 2 groups. Participants in one group will receive the experimental lung plug after the lung biopsy. Participants in the other group will just have the standard lung biopsy without placement of the plug. There is an equal chance of being assigned to either group.

All participants will have the routine lung biopsy performed by their doctor with the aid of a computerized tomography (CT) scan. During a lung biopsy, a needle is inserted into the mass in the lung using the CT for guidance. A smaller needle is then inserted through the first needle to collect a sample of the tissue.

If you are assigned to receive the lung plug, it will be inserted into the track left when the biopsy needle is removed. The smaller sampling needle is removed, and the lung plug is inserted through the larger needle using a delivery tool that has a plunger to push the plug in place. The lung plug remains in the track left when the larger needle is removed.

Regardless of which group you are assigned to, you will be receive the same follow-up treatment. The rates of air leaks after the lung biopsy will be compared between 2 groups of participants. This will provide researchers with the data to learn if the lung plug should be used for all patients receiving a lung biopsy to decrease the number of air leaks.

Your doctor will watch you carefully for air leaks. You will have a chest x-ray about 1 hour after the procedure to again check for air leaks. If a leak is detected, you will receive the normal treatment for air leaks, which includes chest x-rays on a regular basis. If the air leak grows, you may need a chest tube placed for drainage. It is possible that this may require you to stay in the hospital overnight. In the most extreme cases, additional surgery may be needed to stop the air leak. Over time, your body will absorb the plug. A final x-ray will be taken 1 month after the biopsy to be sure that an air leak has not developed.

You will be asked to be in the study for 30 days. This will include the time you spend in the hospital for the biopsy and, if you have an air leak, the entire time you spend in the hospital, if it needs to be treated. In addition, you will return to your doctor the day following the biopsy and 30 days later to have a chest x-ray to look for any late air leaks.

ELIGIBILITY:
Inclusion Criteria:

1. The patient, or legal representative, must understand and provide written consent for the procedure
2. The patient has a non-calcified, radiologically suspicious opacity or lung nodule, including a metastatic lung module, or mass of at least 1.0 cm in size; as determined by CT scan equipped with measurement software. Suspicious nodules observed by CT scan are defined as non-calcified masses with convex borders, not known to be stable. Suspicious nodules can also be defined as masses demonstrating opacity on x-ray that are suspicious by radiographic or clinical means and require biopsy.
3. The patient must meet all medical conditions for lung biopsy;
4. The patient must be at least 18 years of age;

Exclusion Criteria:

1. Patients with radiological findings of bullous emphysema, and the bullae are located near the intended area for biopsy. (Patients may enter the study who have radiological findings of bullous emphysema, as long as the cysts, blebs, or bullae are not in the area of the anticipated biopsy, and biopsy needle track).
2. Female patients who are pregnant. Note: patients of childbearing potential should have a pregnancy test no more than one week prior to the biopsy procedure, and be instructed to have no unprotected sexual intercourse after the test until the biopsy procedure is completed
3. Patients who are uncooperative or cannot follow instructions
4. Patients who are currently enrolled in another Investigational New Drug (IND) or Device Exemption (IDE) clinical investigation that has not completed the required follow-up period
5. Patients who cannot tolerate mild sedation, possibly secondary to poor respiratory status;
6. Patients with fungal infections (Patients with known or imaging evidence highly suggestive of pulmonary fungal infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Gupta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zaetta JM, Licht MO, Fisher JS, Avelar RL; Bio-Seal Study Group. A lung biopsy tract plug for reduction of postbiopsy pneumothorax and other complications: results of a prospective, multicenter, randomized, controlled clinical study. J Vasc Interv Radiol. 2010 Aug;21(8):1235-43.e1-3. doi: 10.1016/j.jvir.2010.04.021. PMID 20656223
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 12, 2005 to February 21, 2008. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: Participants who met the eligibility criteria (77 participants) were consented into study while another set of criteria had to be met for randomization. Only 47 participants met the randomization criteria.
Period: Overall Study
Arm/Group | Pleural Plug | No Pleural Plug
Started | 22 | 25
Completed | 22 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pleural Plug | No Pleural Plug | Total
Number analyzed (Participants) | 22 | 25 | 47
Age Continuous [Median (Full Range); unit: years] | 45 [25 to 85] | 35 [25 to 70] | 45 [25 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absence of Pneumothoraces
Description: Treatment Success defined as absence of pneumothoraces to measure the effects of the hydrogel plug in three follow-up radiographic assessment (x-rays post procedure by 0-60 minutes, 24 hours and 30 days).
Time Frame: X-Rays at 0-60 minutes, 24 hours and 30 days
Population: Intent-to-treat (ITT) population of all subjects who were randomized.
Measure: Number; unit: Participants
Arm/Group | Pleural Plug | No Pleural Plug
Number analyzed (Participants) | 22 | 25
Participants | 18 | 18

ADVERSE EVENTS:
Time Frame: Adverse Event data collected for one year and one month. Adverse Events were documented at 3-timepoints, namely the post-procedure Chest X-Rays (CXRs), 24-hour CXR, and at the 30-day follow up CXR.
Arm/Group | Pleural Plug | No Pleural Plug
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No